CLINICAL TRIAL: NCT02532153
Title: The Impact of Ketamine on the Reward Circuitry of Suicidal Patients: An MRI Study
Brief Title: The Impact of Ketamine on the Reward Circuitry of Suicidal Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No funding.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dawn F Ionescu, Assistant in Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P001783
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Suicidal Ideation; Suicide
Keywords: Suicidal Ideation; Suicide; Suicidal Thoughts; Depression; Ketamine
MeSH Terms: conditions — Suicidal Ideation; Suicide; Depression | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-Label Ketamine (Other)
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Single open-label infusions

SUMMARY:
Every 40 seconds, someone in the world dies by suicide. There is a lack of effective and safe antisuicidal agents for preventing suicide attempts. This leads to the immense worldwide individual, financial, and societal burden of suicide-which is projected to rise in the coming decades-supporting the need for antisuicidal treatments.

This treatment gap may be filled through understanding the neurobiology of suicide, which can guide the development of targeted antisuicidal treatments. Though some research has examined the neurobiology of suicidal ideation in the context of depression-implicating the orbital frontal cortex, anterior cingulate cortex, and striatum-the underlying pathophysiology and neurobiology of suicidal ideation as a separate construct from depression remains largely unknown. Therefore, the investigators propose to study the neurocircuitry of suicidal thoughts, regardless of whether or not depression is present.

ELIGIBILITY:
Inclusion Criteria:

Patients will:

1. be ≥18 years old,
2. read, understand, and provide written informed consent,
3. have suicidal ideation for ≥ 2 months, per the Columbia Suicide Severity Rating Scale (C-SSRS),
4. be on a stable psychiatric medication regimen for ≥28 days,
5. maintain a treating doctor who is in agreement with study participation, and aware of the safety plan in the protocol,
6. have a reliable chaperone accompany them home following the completion of the ketamine infusion day,
7. be generally healthy, as assessed by medical history, physical examination (including vital signs), clinical laboratory evaluations, and electrocardiogram (EKG),
8. be of non-childbearing potential or use of an acceptable form of birth control (females only), and
9. be right handed.

Healthy Controls will:

1. be ≥18 years old,
2. read, understand, and provide written informed consent,
3. have a negative pregnancy test on the morning of the MRI (females only).
4. be right handed.

Exclusion Criteria:

Patients will be excluded if any of the following criteria are met:

1. delirium or dementia diagnosis,
2. unstable medical illness or clinically significant laboratory results,
3. history of clinically significant cardiovascular disease or electrocardiogram (EKG) findings, or medical conditions that put the patient at risk for possible cardiac side effects or alter brain morphology (e.g., diabetes, hypertension, traumatic brain injury), even if well controlled on medications,
4. history of multiple adverse drug reactions,
5. active substance use disorders (except nicotine and caffeine) within the past six months, positive urine toxicology screen, or past history of ketamine/PCP abuse,
6. requirement of excluded medications that may interact with ketamine (e.g., narcotics, barbiturates, sedatives, theophylline, or St. John's Wort),
7. BMI >35,
8. pregnancy, breastfeeding, or unacceptable means of birth control (females only)
9. presence of MRI contraindications (e.g., presence of metallic (ferromagnetic) implants (e.g., heart pacemaker, aneurysm clips)),
10. concurrent participation in other research studies.

Healthy controls will be excluded if any of the following criteria are met:

1. current or past Axis I diagnosis, including alcohol or substance abuse or dependence diagnosis (except for nicotine or caffeine) and suicidal thoughts/attempts,
2. presence of MRI contraindications (e.g., presence of metallic (ferromagnetic) implants (e.g., heart pacemaker, aneurysm clips)),
3. presence of medical illness likely to alter brain morphology and/or physiology (e.g., diabetes) even if controlled by medications,
4. requirement of excluded medications that may interact with ketamine (e.g., narcotics, barbiturates, benzodiazepines, sedatives, theophylline, or St. John's Wort),
5. presence of psychiatric disorders in first-degree relatives,
6. pregnancy, breastfeeding, or unacceptable means of birth control (females only), or
7. BMI >35.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-02 (Estimated); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Columbia Suicide Severity Rating Scale (C-SSRS) | 2 weeks
  Suicide Rating Scale from 1-5; higher numbers indicate increased suicidal thinking

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Ionescu, M.D., Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: MGH Depression Clinical and Research Program — http://www.depressionmgh.org/our-studies